CLINICAL TRIAL: NCT03009890
Title: The Effectiveness of Surgery Versus Casting for Elderly Patients With Displaced Distal Intra-Articular Radius Fractures: A Randomized Controlled Trial
Brief Title: Surgery vs. Casting for Displaced Articular Radius Fractures in Elderly
Acronym: DART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JointResearch (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Maasstad Hospital (Other); Deventer Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL56858.100.16
Record Dates: First submitted 2016-12-22; First posted 2017-01-04 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Radius Distal Fracture
Keywords: elderly; intra articular; RCT
MeSH Terms: conditions — Wrist Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open reduction internal fixation (Experimental): Surgical open reduction internal fixation (ORIF)
  Interventions: Procedure: Surgery (Open Reduction Internal Fixation)
- Plaster immobilization (Active Comparator): Standard local hospital protocol for cast treatment
  Interventions: Procedure: Cast treatment

INTERVENTIONS:
Procedure: Surgery (Open Reduction Internal Fixation) — Either volar of dorsal plating or both
  Other Names: ORIF Open Reduction Internal Fixation
  Arms: Open reduction internal fixation
Procedure: Cast treatment — Hospitals may use their preferred protocol
  Other Names: Plaster
  Arms: Plaster immobilization

SUMMARY:
Objective: to compare the functional outcome after open reduction and internal fixation with non-operative cast treatment for elderly patients with displaced intra-articular distal radius fractures.

DETAILED DESCRIPTION:
Rationale: there is no consensus about the optimal treatment of displaced intra-articular distal radius fractures in elderly patients. To ensure optimal functional outcome there is a tendency to operate. However, there is no evidence that supports the surgical treatment of patients aged 65 years or older and in the absence of clinical trials it stays unclear how elderly patients with intra-articular fractures should be treated.

Study design: multi-center randomized controlled trial with a non-inferiority design. Economic evaluation alongside a randomized controlled multi-center trial.

Study population: all consecutive patients aged between 65 years and older with displaced intra-articular (AO Type C) distal radius fractures, with a not acceptable reduction within 3 weeks following trauma.

Intervention: patients will be randomized between open reduction and internal fixation (intervention group) and plaster immobilization (control group).

Main study parameters: the primary outcome will be evaluated after 1 year with the Patient-Rated Wrist Evaluation score (PRWE). Secondary outcomes comprise other patient reported outcome measures (PROM) including the Disability of the Arm, Shoulder and Hand (DASH), Quality of life (EQ-5D) and Pain Catastrophizing Scale (PCS). Further outcome measurements comprise a costs evaluation questionnaire, range of motion (ROM), grip strength, radiographic parameters and Complications.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years at time of trauma
* Intra-articular distal radius fracture (AO type C*)
* One or more of the following fracture characteristics within 3 weeks post-trauma (including secondary dislocation):

  ≤15° inclination <5 mm radial length >15° dorsal tilt >20° volar tilt intra-articular gap or step-off >2 mm
* < 3 weeks post trauma
* Living independent
* Fit for surgery
* Mentally competent
* Dutch fluency and literacy
* Informed consent

Exclusion Criteria:

* Open fractures
* Neurovascular damage
* Multiple-trauma patients (ISS >16)
* Other fractures in the injured extremity other than ulnar styloid process fractures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
PRWE | 12 months
  Patient-Rated Wrist Evaluation score

SECONDARY OUTCOMES:
DASH | 12 months
  Disability of the Arm, Shoulder and Hand
EQ/5D | 12 months
  Quality of life
PCS | 12 months
  Pain Catastrophizing Scale

OTHER OUTCOMES:
ROM | 12 months
  range of motion
grip strength | 12 months
  grip strength of both wrists
Radiographic parameters | 6 months
  Radial inclination, volar/dorsal tilt, ulnar variance, gap, step off and radial length
Complications | 12 months
  Complications of either treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf W Poolman, Prof. MD PhD, Principal Investigator — OLVG, Amsterdam, the Netherlands
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ter Meulen DP, Mulders MAM, Kruiswijk AA, Kret EJ, Slichter ME, van Dongen JM, Kerkhoffs GMMJ, Goslings JC, Kleinlugtenbelt YV, Willigenburg NW, Schep NWL, Poolman RW; DART Study Group. Effectiveness and cost-effectiveness of surgery versus casting for elderly patients with Displaced intra-Articular type C distal Radius fractures: protocol of a randomised controlled Trial with economic evaluation (the DART study). BMJ Open. 2022 Apr 1;12(4):e051658. doi: 10.1136/bmjopen-2021-051658. PMID 35365511
- See also: website — http://www.dartstudie.nl